CLINICAL TRIAL: NCT00988052
Title: A Multinational, Multicenter, Open-label, Single-assignment Extension of the MS-LAQ-301 (ALLEGRO) Study, to Evaluate the Long-term Safety, Tolerability and Effect on Disease Course of Daily Oral Laquinimod 0.6 mg in Subjects With Relapsing MS
Brief Title: A Study To Evaluate the Long-Term Safety, Tolerability and Effect on Disease Course
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor terminated RRMS studies as sufficient long term clinical data was collected for the study drug in the relevant dose.
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS-LAQ-301E; 2009-012989-30 (EudraCT Number)
Record Dates: First submitted 2009-09-28; First posted 2009-10-01 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Relapsing Multiple Sclerosis
MeSH Terms: interventions — laquinimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Laquinimod (Experimental): One capsule containing 0.6 mg laquinimod to be administered orally once daily.
  Interventions: Drug: Laquinimod

INTERVENTIONS:
Drug: Laquinimod — One capsule containing 0.6 mg laquinimod to be administered orally once daily.

SUMMARY:
The purpose of this study is to make laquinimod 0.6 mg available for all subjects who completed the placebo-controlled MS-LAQ-301 study according to the protocol and to evaluate the long-term safety, tolerability and effect on disease course of daily oral laquinimod 0.6 mg in subjects with relapsing multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have completed the Termination visit of MS-LAQ-301 (completion of all Termination visit activities) according to the MS-LAQ-301 protocol.
2. Women of child-bearing potential must practice an acceptable method of birth control [acceptable methods of birth control in this open label extension phase include: surgical sterilization, intrauterine devices, oral contraceptive, contraceptive patch (or hormone-releasing vaginal ring), long-acting injectable contraceptive, partner's vasectomy or double-barrier method (condom or diaphragm with spermicide)] during the study and up to 30 days after the last dose of the study drug..
3. Subjects must be willing and able to comply with the protocol requirements for the duration of the study.
4. Subjects must be able to comprehend, sign and date a written informed consent prior to entering the MS-LAQ-301E study.

Exclusion Criteria:

1. Premature discontinuation from the MS-LAQ-301 study, for any reason.
2. Pregnancy [according to urine dipstick β-HCG test performed at Baseline (Month 0E) visit] or breastfeeding.
3. Subjects with clinically significant or unstable medical or surgical condition detected or worsened during the MS-LAQ-301 study, which preclude safe participation and completion of the MS-LAQ-301E study. Acute exacerbation of MS will not exclude participation in the MS-LAQ-301E study.
4. Use of inhibitors of CYP3A4 within 2 weeks prior to baseline visit (V0E, Month 0E).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 839 (Actual)
Dates: Start 2009-11-10 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Comi, Prof., MD, Principal Investigator — U.O.Neurology-Neurorehabilitation and Clinical Neurophysiology
Locations (135):
- United States (20):
  - Teva Investigational Site 1076, Phoenix, Arizona
  - Teva Investigational Site 1090, Centennial, Colorado
  - Teva Investigational Site 1088, Fort Collins, Colorado
  - Teva Investigational Site 1102, Northbrook, Illinois
  - Teva Investigational Site 1081, Fort Wayne, Indiana
  - Teva Investigational Site 1083, Des Moines, Iowa
  - Teva Investigational Site 1086, Kansas City, Kansas
  - Teva Investigational Site 1101, Lexington, Kentucky
  - Teva Investigational Site 1096, Farmington Hills, Michigan
  - Teva Investigational Site 1093, Minneapolis, Minnesota
  - Teva Investigational Site 1098, St Louis, Missouri
  - Teva Investigational Site 1082, New York, New York
  - Teva Investigational Site 1073, Winston-Salem, North Carolina
  - Teva Investigational Site 1097, Fargo, North Dakota
  - Teva Investigational Site 1084, Dayton, Ohio
  - Teva Investigational Site 1092, Oklahoma City, Oklahoma
  - Teva Investigational Site 1100, Hershey, Pennsylvania
  - Teva Investigational Site 1075, Lubbock, Texas
  - Teva Investigational Site 1078, San Antonio, Texas
  - Teva Investigational Site 1085, Milwaukee, Wisconsin
- Austria (3):
  - Teva Investigational Site 3300, Klagenfurt
  - Teva Investigational Site 3303, Linz
  - Teva Investigational Site 3302, Sankt Pölten
- Bulgaria (6):
  - Teva Investigational Site 5901, Pleven
  - Teva Investigational Site 5904, Sofia
  - Teva Investigational Site 5903, Sofia
  - Teva Investigational Site 5900, Sofia
  - Teva Investigational Site 5905, Sofia
  - Teva Investigational Site 5902, Varna
- Canada (7):
  - Teva Investigational Site 1132, Bedford, Nova Scotia
  - Teva Investigational Site 1126, London, Ontario
  - Teva Investigational Site 1128, Ottawa, Ontario
  - Teva Investigational Site 1134, Toronto, Ontario
  - Teva Investigational Site 1130, Greenfield Park, Quebec
  - Teva Investigational Site 1129, Montreal, Quebec
  - Teva Investigational Site 1131, Sherbrooke, Quebec
- Czechia (2):
  - Teva Investigational Site 5417, Olomouc
  - Teva Investigational Site 5416, Ostrava - Poruba
- Estonia (2):
  - Teva Investigational Site 5504, Tallinn
  - Teva Investigational Site 5505, Tartu
- France (6):
  - Teva Investigational Site 3525, Besançon
  - Teva Investigational Site 3527, Bron
  - Teva Investigational Site 3526, Clermont-Ferrand
  - Teva Investigational Site 3524, Lille
  - Teva Investigational Site 3528, Marseille
  - Teva Investigational Site 3529, Rennes
- Georgia (2):
  - Teva Investigational Site 8100, Tbilisi
  - Teva Investigational Site 8101, Tbilisi
- Germany (16):
  - Teva Investigational Site 3247, Bayreuth
  - Teva Investigational Site 3241, Berlin
  - Teva Investigational Site 3238, Berlin
  - Teva Investigational Site 3248, Bochum
  - Teva Investigational Site 3245, Dresden
  - Teva Investigational Site 3237, Emden
  - Teva Investigational Site 3242, Erbach im Odenwald
  - Teva Investigational Site 3240, Erfurt
  - Teva Investigational Site 3249, Freiburg im Breisgau
  - Teva Investigational Site 3236, Hamburg
  - Teva Investigational Site 3246, Hamburg
  - Teva Investigational Site 3239, Hanover
  - Teva Investigational Site 3243, Heidelberg
  - Teva Investigational Site 3251, Münster
  - Teva Investigational Site 3250, Trier
  - Teva Investigational Site 3244, Ulm
- Hungary (4):
  - Teva Investigational Site 5115, Budapest
  - Teva Investigational Site 5114, Debrecen
  - Teva Investigational Site 5116, Miskolc
  - Teva Investigational Site 5117, Veszprém
- Israel (4):
  - Teva Investigational Site 8031, Haifa
  - Teva Investigational Site 8030, Jerusalem
  - Teva Investigational Site 8033, Ramat Gan
  - Teva Investigational Site 8032, Tel Aviv
- Italy (9):
  - Teva Investigational Site 3044, Catania
  - Teva Investigational Site 3045, Fidenza
  - Teva Investigational Site 3042, Gallarate
  - Teva Investigational Site 3046, Grosseto
  - Teva Investigational Site 3038, Milan
  - Teva Investigational Site 555, Milan
  - Teva Investigational Site 3039, Milan
  - Teva Investigational Site 3041, Palermo
  - Teva Investigational Site 3040, Rome
- Lithuania (2):
  - Teva Investigational Site 5704, Kaunas
  - Teva Investigational Site 5705, Šiauliai
- Netherlands (2):
  - Teva Investigational Site 3810, Nieuwegein
  - Teva Investigational Site 3809, Nijmegen
- Poland (8):
  - Teva Investigational Site 5322, Częstochowa
  - Teva Investigational Site 5319, Gmina Końskie
  - Teva Investigational Site 5320, Gorzów Wielkopolski
  - Teva Investigational Site 5316, Katowice
  - Teva Investigational Site 5318, Kielce
  - Teva Investigational Site 5317, Krakow
  - Teva Investigational Site 5315, Lodz
  - Teva Investigational Site 5325, Warsaw
- Romania (5):
  - Teva Investigational Site 5208, Bucharest
  - Teva Investigational Site 5210, Cluj-Napoca
  - Teva Investigational Site 5212, Constanța
  - Teva Investigational Site 5211, Târgu Mureş
  - Teva Investigational Site 5209, Timișoara
- Russia (10):
  - Teva Investigational Site 5021, Moscow
  - Teva Investigational Site 5028, Nizhny Novgorod
  - Teva Investigational Site 5027, Novosibirsk
  - Teva Investigational Site 5030, Perm
  - Teva Investigational Site 5026, Saint Petersburg
  - Teva Investigational Site 5025, Saint Petersburg
  - Teva Investigational Site 5024, Saint Petersburg
  - Teva Investigational Site 5022, Saint Petersburg
  - Teva Investigational Site 5023, Saint Petersburg
  - Teva Investigational Site 5029, Yekaterinburg
- Serbia (2):
  - Teva Investigational Site 6100, Belgrade
  - Teva Investigational Site 6102, Niš
- Spain (13):
  - Teva Investigational Site 3132, Barcelona
  - Teva Investigational Site 3134, Barcelona
  - Teva Investigational Site 3144, Barcelona
  - Teva Investigational Site 3140, Beade-Pontevedra
  - Teva Investigational Site 3142, Getafe
  - Teva Investigational Site 3135, Lleida
  - Teva Investigational Site 3133, Madrid
  - Teva Investigational Site 3146, Madrid
  - Teva Investigational Site 3137, Murcia
  - Teva Investigational Site 3138, Pontevedra
  - Teva Investigational Site 3136, Salt
  - Teva Investigational Site 3139, Santiago de Compostela
  - Teva Investigational Site 3143, Valencia
- Sweden (3):
  - Teva Investigational Site 4204, Stockholm
  - Teva Investigational Site 4205, Stockholm
  - Teva Investigational Site 4206, Stockholm
- Teva Investigational Site 8201, Izmir, Turkey (Türkiye)
- Ukraine (5):
  - Teva Investigational Site 5803, Dnipropetrovsk
  - Teva Investigational Site 5802, Kyiv
  - Teva Investigational Site 5804, Kyiv
  - Teva Investigational Site 5800, Lviv
  - Teva Investigational Site 5801, Vinnytsia
- United Kingdom (3):
  - Teva Investigational Site 3425, Liverpool
  - Teva Investigational Site 3424, London
  - Teva Investigational Site 3422, Sheffield

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the preceding double-blind, placebo-controlled ALLEGRO study (study MS-LAQ-301), 1106 subjects with RRMS were randomized to treatment, and 864 subjects completed the study according to the protocol (ie, by completing the ALLEGRO study termination visit procedures).
Pre-assignment Details: In this open-label extension study, 839 subjects with RRMS were enrolled to receive laquinimod 0.6 mg at 135 study sites in 22 countries by 135 investigators.
Groups:
- Early Laquinimod: All participants in MS-LAQ-301E were administered 1 capsule containing laquinimod 0.6 mg taken orally at the same hour every day until the product was commercially available or development stopped.
  The Early laquinimod subgroup included participants in MS-LAQ-301 double-blind study who were administered laquinimod 0.6 mg daily for 24 months.
- Switch From Placebo: All participants in MS-LAQ-301E were administered 1 capsule containing laquinimod 0.6 mg taken orally at the same hour every day until the product was commercially available or development stopped.
  The Switch from placebo subgroup included participants in MS-LAQ-301 double-blind study who were administered placebo daily for 24 months.
Period: Overall Study
Arm/Group | Early Laquinimod | Switch From Placebo
Started | 423 | 416
Completed | 0 | 0
Not Completed | 423 | 416
Not completed — Missing | 1 | 0
Not completed — Teva requested subject withdrawal | 3 | 1
Not completed — Death | 1 | 3
Not completed — Protocol Violation | 6 | 5
Not completed — Pregnancy | 6 | 6
Not completed — Lack of Efficacy | 8 | 7
Not completed — Lost to Follow-up | 6 | 11
Not completed — Physician Decision | 27 | 28
Not completed — Adverse Event | 35 | 28
Not completed — Withdrawal by Subject | 90 | 91
Not completed — Study terminated by sponsor | 240 | 236

BASELINE CHARACTERISTICS:
Population: Participants enrolled in the MS-LAQ-301 extension study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Laquinimod | Switch From Placebo | Total
Number analyzed (Participants) | 423 | 416 | 839
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (9.10) | 40.5 (9.14) | 40.8 (9.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 298 | 271 | 569
  Male | 125 | 145 | 270
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian / Oriental | 2 | 0 | 2
  Black / African American | 1 | 5 | 6
  Caucasian | 414 | 401 | 815
  Other | 2 | 2 | 4
  Missing | 1 | 2 | 3
  Unknown | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A treatment-emergent adverse event was defined as any untoward medical occurrence that develops or worsens in severity following start of treatment and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents normal daily activities. Relation of AE to treatment was determined by the investigator. Serious AEs (SAE) include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes. TEAEs associated with cancer, ischemic heart disease, cerebrovascular events, and arthritis were considered to be of special interest.
Time Frame: Day 1 up to 7.64 years
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Early Laquinimod | Switch From Placebo
Number analyzed (Participants) | 423 | 416
Participants
  =>1 TEAE | 375 | 374
  =>1 Severe TEAE | 76 | 69
  =>1 TEAE of special interest | 109 | 105
  =>1 treatment-related TEAE | 139 | 153
  =>1 TEAE leading to death | 3 | 3
  =>1 Serious TEAE | 108 | 92
  =>1 TEAE causing discontinuation | 35 | 32

2. Secondary Outcome: Participants With Potentially Clinically Significant Abnormal Vital Signs
Description: Vital signs with potentially clinically significant abnormal results were evaluated using the following significance criteria:
  * Pulse rate low: <=45 and decrease >=30 beats/minute
  * Pulse rate high: >=120 and increase >=30 beats/minute
  * Systolic blood pressure low: <=90 and decrease >=30 mmHg
  * Systolic blood pressure high: >=180 and increase >=30 mmHg
  * Diastolic blood pressure low: <=50 and decrease >=20 mmHg
  * Diastolic blood pressure high: >=100 and increase >=20 mmHg
Time Frame: Day 1 up to 7.64 years
Population: Safety analysis set of participants with a baseline and post-baseline value for that vital sign.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Laquinimod | Switch From Placebo
Number analyzed (Participants) | 423 | 416
Participants
  Participants with at least one abnormality | 36 | 34
  Pulse rate - low | 1 | 1
  Pulse rate - high | 2 | 1
  Systolic blood pressure - low | 20 | 10
  Systolic blood pressure - high | 1 | 2
  Diastolic blood pressure - low | 7 | 7
  Diastolic blood pressure - high | 8 | 14

3. Secondary Outcome: Participants With Serum Chemistry Laboratory Tests That Were Potentially Clinically Significant (PCS) Abnormal Comparing Baseline to Any Time During the Study
Description: Counts include two conditions:
  * a change from High / Non-PCS at baseline to Low PCS at any point during the study
  * a change from Low / Non-PCS at baseline to High PCS at any point during the study Participants whose condition was not changed from baseline or was changed to a non- PCS value are included in the population count. ALT=alanine aminotransferase ALP=alkaline phosphatase P-amylase=amylase, pancreatic AST=aspartate aminotransferase CRP=C reactive protein CK=creatine kinase CTN=creatinine FIB=fibrinogen GGT=gamma glutamyl transferase K=potassium
Time Frame: Day 1 up to 7.64 years
Population: Safety analysis set of participants with both a baseline and a post-baseline value for the test.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Laquinimod | Switch From Placebo
Number analyzed (Participants) | 422 | 415
Participants
  ALT - change from Low / Non- PCS to High PCS | 8 | 14
  Albumen - change from High / Non-PCS to Low PCS | 1 | 0
  ALP - change from Low / Non- PCS to High PCS | 3 | 0
  p-Amylase - change from Low / Non-PCS to High PCS | 2 | 6
  AST - change from Low / Non- PCS to High PCS | 4 | 5
  CRP - change from Low / Non- PCS to High PCS | 41 | 51
  Calcium - change from High / Non-PCS to Low PCS | 1 | 4
  Calcium - change from Low / Non-PCS to High PCS | 1 | 2
  CK - change from Low / Non- PCS to High PCS | 16 | 17
  CTN - change from Low / Non- PCS to High PCS | 2 | 2
  FIB - change from Low / Non- PCS to High PCS | 37 | 38
  GGT - change from Low / Non- PCS to High PCS | 33 | 24
  Glucose - change from High / Non-PCS to Low PCS | 23 | 27
  Glucose - change from Low / Non-PCS to High PCS | 9 | 5
  Phosphate-change from High / Non-PCS to Low PCS | 14 | 15
  Phosphate-change from Low / Non-PCS to High PCS | 19 | 16
  K - change from High / Non- PCS to Low PCS | 4 | 3
  K - change from Low / Non- PCS to High PCS | 46 | 55
  Sodium - change from High / Non-PCS to Low PCS | 8 | 3
  Sodium - change from Low / Non-PCS to High PCS | 13 | 17
  Urea - change from Low / Non- PCS to High PCS | 3 | 4

4. Secondary Outcome: Participants With Serum Hematology Laboratory Tests That Were Potentially Clinically Significant (PCS) Abnormal Comparing Baseline to Any Time During the Study
Description: Counts include two conditions:
  * a change from High / Non-PCS at baseline to Low PCS at any point during the study
  * a change from Low / Non-PCS at baseline to High PCS at any point during the study Participants whose condition was not changed from baseline or was changed to a non- PCS value are included in the population count.
Time Frame: Day 1 up to 7.64 years
Population: Safety analysis set of participants with both a baseline and a post-baseline value for the test.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Laquinimod | Switch From Placebo
Number analyzed (Participants) | 422 | 415
Participants
  Hematocrit - change from High / Non-PCS to Low PCS | 36 | 29
  Hemoglobin -change from High / Non-PCS to Low PCS | 27 | 22
  Hemoglobin -change from Low / Non-PCS to High PCS | 0 | 1
  Leukocytes - change from High / Non-PCS to Low PCS | 1 | 1
  Leukocytes - change from Low / Non-PCS to High PCS | 4 | 3
  Neutrophils - change from High/Non-PCS to Low PCS | 15 | 12
  Platelets - change from High / Non-PCS to Low PCS | 4 | 7
  Platelets - change from Low / Non-PCS to High PCS | 2 | 6

5. Secondary Outcome: Participants With Electrocardiogram (ECG) Fiindings That Shifted From Baseline to Any Time During the Study
Description: Shifts are presented as Baseline finding / Worse finding at anytime during the study.
  Categories for findings are:
  * normal
  * abnormal, not clinically significant (Not CS)
  * abnormal, clinically significant (CS)
Time Frame: Day 1 up to 7.64 years
Population: Safety analysis set of participants with both a baseline and a post-baseline ECG.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Laquinimod | Switch From Placebo
Number analyzed (Participants) | 420 | 412
Participants
  Normal / Normal | 189 | 198
  Normal / Abnormal, Not CS | 145 | 126
  Normal / Abnormal, CS | 2 | 3
  Abnormal, Not CS / Normal | 12 | 14
  Abnormal, Not CS / Abnormal, Not CS | 70 | 67
  Abnormal, Not CS / Abnormal, CS | 2 | 4
  Abnormal, CS / Normal | 0 | 0
  Abnormal, CS / Abnormal, Not CS | 0 | 0
  Abnormal, CS / Abnormal, CS | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to 7.64 years
Groups:
- Early Laquinimod 0.6 mg: All participants in MS-LAQ-301E were administered 1 capsule containing laquinimod 0.6 mg taken orally at the same hour every day until the product was commercially available or development stopped.
  The Early laquinimod subgroup included participants in MS-LAQ-301 double-blind study who were administered laquinimod 0.6 mg daily for 24 months.
- Switch From Placebo to Laquinimod 0.6 mg: All participants in MS-LAQ-301E were administered 1 capsule containing laquinimod 0.6 mg taken orally at the same hour every day until the product was commercially available or development stopped.
  The Switch from placebo subgroup included participants in MS-LAQ-301 double-blind study who were administered placebo daily for 24 months.
Arm/Group | Early Laquinimod 0.6 mg | Switch From Placebo to Laquinimod 0.6 mg
All-Cause Mortality (participants affected / at risk) | 3/423 | 3/416
Serious Adverse Events (participants affected / at risk) | 108/423 | 92/416
Other Adverse Events (participants affected / at risk) | 299/423 | 300/416
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Laquinimod 0.6 mg (N=423) | Switch From Placebo to Laquinimod 0.6 mg (N=416)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Bone marrow oedema (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Silent myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0)
Parathyroid gland enlargement (Endocrine disorders) | 1 (1) | 0 (0)
Blindness unilateral (Eye disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Omental infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Drowning (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Medical device pain (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hydrocholecystis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 4 (4) | 3 (3)
Appendicitis perforated (Infections and infestations) | 2 (2) | 1 (1)
Bartholin's abscess (Infections and infestations) | 1 (2) | 0 (0)
Breast abscess (Infections and infestations) | 1 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 2 (2) | 0 (0)
Hepatic echinococciasis (Infections and infestations) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Latent syphilis (Infections and infestations) | 1 (1) | 0 (0)
Latent tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (2)
Mycotoxicosis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0)
Ovarian abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 4 (4) | 0 (0)
Periumbilical abscess (Infections and infestations) | 1 (1) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (4)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 1 (1)
Salpingo-oophoritis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 4 (4) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Joint instability (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Knee impingement syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendon calcification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia stage 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Langerhans' cell histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tubular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (2)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 3 (3) | 2 (2)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Simple partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (3)
Agoraphobia (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Mood disorder due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0)
Neurosis (Psychiatric disorders) | 1 (1) | 0 (0)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Bladder dysfunction (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Ketonuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral meatus stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Acquired hydrocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (2) | 2 (2)
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hydrosalpinx (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pharyngeal polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Intervertebral disc operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Laquinimod 0.6 mg (N=423) | Switch From Placebo to Laquinimod 0.6 mg (N=416)
Anaemia (Blood and lymphatic system disorders) | 22 (25) | 16 (17)
Abdominal pain upper (Gastrointestinal disorders) | 19 (23) | 31 (39)
Diarrhoea (Gastrointestinal disorders) | 24 (31) | 21 (23)
Nausea (Gastrointestinal disorders) | 24 (27) | 26 (37)
Fatigue (General disorders) | 25 (30) | 31 (38)
Bronchitis (Infections and infestations) | 33 (44) | 33 (46)
Influenza (Infections and infestations) | 28 (41) | 34 (46)
Nasopharyngitis (Infections and infestations) | 106 (169) | 112 (210)
Sinusitis (Infections and infestations) | 27 (36) | 28 (47)
Upper respiratory tract infection (Infections and infestations) | 43 (69) | 41 (65)
Urinary tract infection (Infections and infestations) | 55 (110) | 39 (76)
Fall (Injury, poisoning and procedural complications) | 20 (30) | 23 (30)
Alanine aminotransferase increased (Investigations) | 13 (16) | 22 (27)
C-reactive protein increased (Investigations) | 26 (31) | 31 (37)
Gamma-glutamyltransferase increased (Investigations) | 22 (27) | 16 (23)
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 (57) | 47 (59)
Back pain (Musculoskeletal and connective tissue disorders) | 78 (127) | 77 (124)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 (15) | 25 (29)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 (35) | 33 (45)
Headache (Nervous system disorders) | 57 (132) | 86 (160)
Multiple sclerosis relapse (Nervous system disorders) | 17 (35) | 29 (36)
Depression (Psychiatric disorders) | 35 (41) | 28 (35)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (26) | 35 (40)
Hypertension (Vascular disorders) | 32 (32) | 26 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT00988052/Prot_SAP_000.pdf